CLINICAL TRIAL: NCT00902343
Title: A Prospective Randomized Controlled Trial Comparing Nomogram-based Versus Standard Allocation of Acute Normovolemic Hemodilution (ANH) During Hepatic Resection
Brief Title: Controlled Trial Comparing Nomogram-based Versus Standard Allocation of Acute Normovolemic Hemodilution (ANH) During Hepatic Resection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-158
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Liver Cancer
Keywords: Liver; Cancer; Primary; Metastatic; transfusions; 08-158
MeSH Terms: conditions — Liver Neoplasms; Neoplasms; Neoplasm Metastasis

ARMS (2):
- 1 (Experimental): nomogram-based selection for acute normovolemic hemodilution
  Interventions: Procedure: nomogram-based selection for acute normovolemic hemodilution
- 2 (Active Comparator): standard selection for ANH based on a planned resection of 3 or more segments.
  Interventions: Procedure: standard selection for ANH based on a planned resection of 3 or more segments

INTERVENTIONS:
Procedure: nomogram-based selection for acute normovolemic hemodilution — Will use the nomogram to determine whether or not the patient needs ANH during surgery. The nomogram assigns a point value to certain pre-op factors to determine whether or not the patient will need an ANH. Preoperative factors that will be used are platelet count, planned amount of liver to be removed, hemoglobin level, if the surgeon needs to operate on any organ outside of the liver to remove the tumor, and the patients health overall.
  Other Names: The actual operation to remove the tumor will be the same for both groups,; and in fact will be done the same way as it is done for patients who are not; in this study.
  Arms: 1
Procedure: standard selection for ANH based on a planned resection of 3 or more segments — Will use the planned amount of liver to be removed to determine whether or not the patient needs an ANH during surgery.
  Other Names: The actual operation to remove the tumor will be the same for both groups,; and in fact will be done the same way as it is done for patients who are not; in this study.
  Arms: 2

SUMMARY:
The purpose of this study is to learn the best method of assigning patients to receive "acute normovolemic hemodilution" during liver surgery.

DETAILED DESCRIPTION:
For many patients, the best treatment for tumors in the liver is surgery, which is called liver resection. With major liver surgery, there is a chance that you will require a transfusion of blood products (either red blood cells or plasma) either during, or a few days after surgery. The surgeons at Memorial Sloan-Kettering Cancer Center (MSKCC) perform a very large number of liver resections every year, and have pioneered techniques that minimize bleeding during the operation. Even so, liver operations such as the one you will undergo have a 30% chance of requiring a transfusion. One technique that has been shown to lower the need for transfusions is called "acute normovolemic hemodilution (ANH)". ANH was first introduced over 20 years ago, and has been used in many types of operations, including liver resection. The studies done on ANH here at MSKCC and at other hospitals suggest that it may help conserve blood and lower the risk of you needing a blood transfusion. In fact, a recent study completed here showed that patients who received ANH while undergoing a major liver resection were half as likely to require a blood transfusion.

Researchers at MSKCC are conducting a study to determine the best way to assign patients to receive ANH. Currently, patients are assigned to undergo ANH based on the amount of liver that is expected to be removed (also called 'extent of resection'). We are looking at whether assigning patients to receive ANH based on a nomogram more appropriately selects patients who would benefit from undergoing ANH. A nomogram is a predictive mathematical tool that uses a point system to evaluate each patient's anticipated blood transfusion needs based on the data from many previous patients with the same condition(s). Using this method, your risk of requiring a blood transfusion will be calculated, and depending on the predicted risk of transfusion, you may or may not be selected to undergo ANH. All patients will undergo randomization (a computer-generated decision, as in the flip of a coin): half will be assigned to the arm using the nomogram-based selection for ANH, and half will be assigned based on the planned operative procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years).
* Preoperative hemoglobin concentration ≥ 11 mg/dl (males), ≥ 10 mg/dl (females) within 14 days of registration.
* Patients scheduled for hepatic resection for any indication, with or without other planned procedures

Exclusion Criteria:

* A history of active coronary artery disease.
* Patients with a history of coronary artery disease will be eligible if they have had a cardiac stress study showing no reversible ischemia and normal LV function within 30 days of operation.
* Patients with active or symptomatic cerebrovascular disease; patients with hemodynamically insignificant stenosis will not be deemed ineligible.
* A history of congestive heart failure.
* A history of uncontrolled hypertension.
* A history of restrictive or obstructive pulmonary disease.
* A history of renal dysfunction (Cr > 1.8).
* Abnormal coagulation parameters (INR > 1.5 in patients not on coumadin; an INR>1.5 is acceptable in patients still on coumadin, provided drug is discontinued no less than 4 days prior to operation.)
* Presence of active infection.
* Evidence of hepatic metabolic disorder (bilirubin > 2 mg/dl, ALT > 75 U/L in the absence of biliary tract obstruction).
* Pre-operative autologous blood donation.
* Erythropoietin use
* Patients scheduled for ablation only
* Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2009-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
To determine if nomogram-based allocation of ANH is superior to allocation using extent of resection alone (planned resection of 3 or more liver segments) in patients undergoing partial hepatectomy. | during surgery

SECONDARY OUTCOMES:
To assess the impact of nomogram-based allocation of ANH compared to standard allocation on the need for fresh frozen plasma (FFP) transfusions. | during surgery

CONTACTS AND LOCATIONS:
Overall Officials: William Jarnagin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm